CLINICAL TRIAL: NCT03450590
Title: Relation Between Heart Rate Variability and Cardiorespiratory Complications During Ophthalmic Arterial Chemotherapy for Retinoblastoma
Brief Title: Heart Rate Variability and Cardiorespiratory Complications During Ophthalmic Arterial Chemotherapy for Retinoblastoma
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Tae Kyong Kim, Clinical assistant professor, Seoul National University Hospital
Other Study IDs: IAchemo_HRV
Record Dates: First submitted 2018-02-22; First posted 2018-03-01 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-10

CONDITIONS: Parasympathetic Cardiovascular Function Disorder
Keywords: heart rate variability; intraarterial chemotherapy; ophthalmic arterial chemotherapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A patient undergoing ophthalmic arterial chemosurgery may experience a sudden, profound decrease in lung compliance when the microcatheter is in the ICA or ophthalmic artery. However, underlying pathophysiology of the respiratory complication is unknown. In this study, the investigators are going to investigate the relation between underlying balance of parasympathetic and sympathetic tone and the respiratory complications by analyzing heart rate beat-to-beat variability.

DETAILED DESCRIPTION:
A patient undergoing ophthalmic arterial chemosurgery may experience a sudden, profound decrease in lung compliance when the microcatheter is in the ICA or ophthalmic artery. However, underlying pathophysiology of the respiratory complication is unknown. In this study, the investigators are going to investigate the relation between underlying balance of parasympathetic and sympathetic tone and the respiratory complications by analyzing heart rate beat-to-beat variability. Also, the investigators are going to investigate whether baseline heart rate variability can predict respiratory complications during the procedures.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing ophthalmic arterial chemotherapy

Exclusion Criteria:

* None

Max Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients undergoing ophthalmic arterial chemotherapy for retinoblastoma
Sampling Method: Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2019-09-09 (Actual); Study Completion 2019-09-09 (Actual)

PRIMARY OUTCOMES:
Heart rate variability | 5 min after microcatheter enters ophthalmic artery
  Heart rate variability

SECONDARY OUTCOMES:
Heart rate variability | 5 min after anesthesia induction
  Heart rate variability
Heart rate variability | 5 min before end of anesthesia
  Heart rate variability

CONTACTS AND LOCATIONS:
Overall Officials: Tae Kyong Kim, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea